CLINICAL TRIAL: NCT03666845
Title: Plasma Ropivacaine Concentrations After Peripheral Nerve Block in Patients With Severe Renal Dysfunction
Brief Title: Plasma Ropivacaine Concentrations After Sciatic Nerve Block in Patients With Chronic Kidney Disease
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor, Seoul National University Hospital
Other Study IDs: H-1807-153-961
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Regional Anesthesia Morbidity; Local Anesthetic Drug Adverse Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Arterial blood sampling will be taken at 2.5, 5, 15, 30, 60 minutes and 2, 6, 24 hours after sciatic nerve block.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sciatic nerve block: Patients scheduled for foot and ankle surgery under sciatic nerve block and who had chronic kidney disease
  Interventions: Procedure: Sciatic nerve block

INTERVENTIONS:
Procedure: Sciatic nerve block — Sciatic nerve block will be performed using ropivacaine (2.5mg/kg) under ultrasound-guidance with nerve stimulator.
  Other Names: Popliteal block

SUMMARY:
This prospective observational study aimed to examine the pharmacokinetics of ropivacaine in patients with chronic kidney disease after sciatic nerve block.

Sciatic nerve block for foot and ankle surgery will be performed using ropivacaine under ultrasound-guidance, and arterial blood test will be taken for total plasma ropivacaine concentration at 2.5, 5, 15, 30, 60 minutes and 2, 6, 24 hours after sciatic nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for foot and ankle surgery
* Patients with chronic kidney disease (glomerular filtration rate < 60 ml/min/1.73m2) (changed from 30 ml/min/1.73m2 to facilitate patient recruitment)
* Patients who are thought to be clinically helpful to receive sciatic nerve block rather than general anesthesia because of comorbidities such as cardiopulmonary dysfunction and cerebral dysfunction

Exclusion Criteria:

* Patients who need to renal replacement therapy, such as hemodialysis
* Patients with liver disease (aspartate transaminase OR alanine transaminase > 80 IU/L)
* Patients with allergic disease
* Patients with previous history of drug allery
* Patients with chronic pain persisting 3 months

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for foot and ankle surgery under sciatic nerve block and who had chronic kidney disease
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2023-12-28 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of unbound ropivacaine | 2.5, 5, 15, 30, 60 minutes and 2, 6, 24 hours after sciatic nerve block
  whether the unbound plasma concentration of ropivacaine was maintained under 0.56 mcg/ml that was determined as toxic level in a previous study.

SECONDARY OUTCOMES:
Plasma concentration of 3-OH-ropivacaine | 2.5, 5, 15, 30, 60 minutes and 2, 6, 24 hours after sciatic nerve block
  metabolite of ropivacaine
Plasma concentration of pipecoloxylidide | 2.5, 5, 15, 30, 60 minutes and 2, 6, 24 hours after sciatic nerve block
  metabolite of ropivacaine
Postoperative pain score | 2, 6, 24 hours after sciatic nerve block
  11-point numeric rating scale ranging from '0' representing one extreme (e.g. "extremely dissatisfied") to '10' representing the other extreme (e.g. "extremely satisfied")
Local anesthetic systemic toxicity | 2, 6, 24 hours after sciatic nerve block
  numbness of the tongue, twitching, convulsion, dysarrhythmia, coma

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, Pf., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea